CLINICAL TRIAL: NCT05345860
Title: Adopting the MRD Strategy to Optimize Post-operation Adjuvant Therapies for Early Stage Breast Cancer, a Prospective Cohort Study
Brief Title: Adopting the MRD Strategy to Optimize Post-operation Adjuvant Therapies for Early Stage Breast Cancer
Acronym: AMENDER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Huanxing Cancer Hospital (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Deputy Director of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC3397
Record Dates: First submitted 2022-04-18; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Early-stage Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- TNBC with high risk or MRD+ (Experimental): TNBC patients with clinical high risk or post-operation 1st MRD tested positive.
  It's possible that this arm will be divided into many sub-arms considering the different kinds of intensive adjuvant therapies and the adopting of MRD strategy.
  Interventions: Other: The MRD strategy for high risk or MRD+ TNBC patients
- HER2+ with high risk or MRD+ (Experimental): HER2+ patients with clinical high risk or post-operation 1st MRD tested positive.
  It's possible that this arm will be divided into many sub-arms considering the different kinds of intensive adjuvant therapies and the adopting of MRD strategy.
  Interventions: Other: The MRD strategy for high risk or MRD+ HER2+ patients
- ER+ with high risk or MRD+ (Experimental): ER+ patients with clinical high risk or post-operation 1st MRD tested positive.
  It's possible that this arm will be divided into many sub-arms considering the different kinds of intensive adjuvant therapies and the adopting of MRD strategy.
  Interventions: Other: The MRD strategy for high risk or MRD+ ER+ patients
- TNBC with low risk and MRD- (Experimental): TNBC patients with low clinical risk and post-operation 1st MRD tested negative.
  It's possible that this arm will be divided into many sub-arms considering the different kinds of standard adjuvant therapies and the adopting of MRD strategy.
  Interventions: Other: The MRD strategy for low risk and MRD- TNBC patients
- HER2+ with low risk and MRD- (Experimental): HER2+ patients with low clinical risk and post-operation 1st MRD tested negative.
  It's possible that this arm will be divided into many sub-arms considering the different kinds of standard adjuvant therapies and the adopting of MRD strategy.
  Interventions: Other: The MRD strategy for low risk and MRD- HER2+ patients
- ER+ with low risk and MRD- (Experimental): ER+ patients with low clinical risk and post-operation 1st MRD tested negative.
  It's possible that this arm will be divided into many sub-arms considering the different kinds of standard adjuvant therapies and the adopting of MRD strategy.
  Interventions: Other: The MRD strategy for low risk and MRD- ER+ patients

INTERVENTIONS:
Other: The MRD strategy for high risk or MRD+ TNBC patients — Standard adjuvant chemotherapy + additional chemotherapy:
  * BRCA positive patients: standard adjuvant chemotherapy + olaparib
  * BRCA negative patients: standard adjuvant chemotherapy + capecitabine
  In the period of once 3 months follow-up, if MRD remains positive, the additional chemotherapy will be changed for at most once.
  Arms: TNBC with high risk or MRD+
Other: The MRD strategy for high risk or MRD+ HER2+ patients — Standard adjuvant chemotherapy + intensive targeted therapy:
  * Neoadjuvant therapy non-pCR patients: standard adjuvant chemotherapy completed+ T-DM1/HP
  * Neoadjuvant therapy pCR patients: standard adjuvant chemotherapy completed + HP
  * Adjuvant therapy patients: AC-T/TCb + HP
  In the period of once 3 months follow-up, if MRD remains positive, the intensive targeted therapy will be changed for at most once.
  Arms: HER2+ with high risk or MRD+
Other: The MRD strategy for high risk or MRD+ ER+ patients — Standard adjuvant chemotherapy + intensive endocrine therapy:
  * Premenopausal patients: Standard adjuvant chemotherapy followed by OFS + TAM/TOR, OFS + ANA/LET/EXE, or OFS + ANA/LET/EXE + Abemaciclib.
  * Postmenopausal: Standard adjuvant chemotherapy followed by ANA/LET/EXE + Abemaciclib.
  In the period of once 3 months follow-up, if MRD remains positive, the intensive endocrine therapy will be changed for at most once.
  Arms: ER+ with high risk or MRD+
Other: The MRD strategy for low risk and MRD- TNBC patients — Standard adjuvant chemotherapy: AC-T/TC/TCb/AC.
  In the period of once 3 months follow-up, if MRD turns positive, additional adjuvant therapies listed in "The MRD strategy for high risk or MRD+ TNBC patients "will be added for at most twice.
  Arms: TNBC with low risk and MRD-
Other: The MRD strategy for low risk and MRD- HER2+ patients — Standard adjuvant chemotherapy + standard targeted therapy:
  * Neoadjuvant therapy pCR patients: standard adjuvant chemotherapy (AC-T/TC/TCb) completed + H.
  * Adjuvant therapy patients: AC-T/TC/TCb/wP + H.
  In the period of once 3 months follow-up, if MRD turns positive, additional adjuvant targeted therapies listed in "The MRD strategy for high risk or MRD+ HER2+ patients "will be added for at most twice.
  Arms: HER2+ with low risk and MRD-
Other: The MRD strategy for low risk and MRD- ER+ patients — Standard adjuvant chemotherapy + standard endocrine therapy:
  * Premenopausal patients: Standard adjuvant chemotherapy followed by TAM/TOR.
  * Postmenopausal patients: Standard adjuvant chemotherapy followed by ANA/LET/EXE.
  In the period of once 3 months follow-up, if MRD turns positive, additional adjuvant endocrine therapies listed in "The MRD strategy for high risk or MRD+ ER+ patients "will be added for at most twice.
  Arms: ER+ with low risk and MRD-

SUMMARY:
This study is a prospective, multi-center, open-label cohort study, with 3 years disease free survival(DFS) as the primary endpoint. We optimize post-operation adjuvant therapy for early stage breast cancer based on the MRD strategy: patients with clinical high risk or post-operation 1st MRD tested positive will receive intensive adjuvant therapy, while patients with low clinical risk and post-operation 1st MRD tested negative will receive standard adjuvant therapy, and the treatment regimens will be adjusted every 3 months according to the change of MRD status. About 100 TNBC patients, 100 HER2+ patients, and 100 ER+ patients are planned to be enrolled.

DETAILED DESCRIPTION:
MRD will be tested with tumor-informed personalized panel in this trail. The adjuvant therapies in the MRD strategy are all standard therapies in guidelines of China or abroad.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥18 years (inclusive).
* Histologically confirmed, perioperative invasive breast cancer that is resectable without metastasis(stage I-III).
* No anti-breast cancer systematic therapy received, and planning to receive surgery and systemic therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* With Adequate Organ Function:

  a. Bone marrow function: Hemoglobin ≥ 10 g/dL; Absolute leucocyte count ≥ 4×10^9/L; Absolute neutrophil count ≥ 1.5×10^9/L; Platelets ≥ 100 × 10^9/L; b. Liver function (based on the normal values specified by study site): Serum total bilirubin ≤ 1.5 × the upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; c. Renal function (based on the normal values specified by study site): Serum creatinine ≤ 1.5 × ULN.
* The patients voluntarily signed an informed consent form.

Exclusion Criteria:

* Known to have other aggressive malignant tumor that is progressing or requires systemic treatment in the past 5 years (does not exclude subjects with skin basal cell carcinoma, skin squamous cell carcinoma, breast ductal carcinoma in situ or cervical cancer in situ that has received curative treatment).
* Have a clear history of neurological or mental disorders, including epilepsy or dementia, etc.; have a history of psychotropic drug abuse or drug abuse.
* Known history of allergy to the drug components in MRD strategy; history of immunodeficiency, or history of organ transplantation.
* There are other concomitant diseases that seriously threaten the patient's safety or affect the patient's completion of the study, such as serious infection, liver disease, cardiovascular disease, kidney disease, respiratory disease or uncontrolled diabetes or dyslipidemia.
* Female patients during pregnancy or lactation.
* The investigator determines that subjects are not appropriate to participate in the study due to other factors.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-03-24 (Estimated); Study Completion 2027-03-24 (Estimated)

PRIMARY OUTCOMES:
3 years disease free survival(DFS) | From date of radical surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  the period after curative treatment [disease eliminated] when no disease can be detected

SECONDARY OUTCOMES:
5 years disease free survival(DFS) | From date of radical surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  the period after curative treatment [disease eliminated] when no disease can be detected
1 years disease free survival(DFS) | From date of radical surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  the period after curative treatment [disease eliminated] when no disease can be detected
Overall Survival(OS) | From date of radical surgery until the date of death from any cause, assessed up to 60 months
  OS was defined as the time from the date of radical surgery to the date of death from any cause
Adverse events (AEs) | Up to 5 years
  The drug safety was assessed by investigator(s) according to NCI-CTCAE v5.0.
quality of life (QoL) | Up to 5 years
  QoL measurement is conducted in the hospital after treatment via digital questionnaire EORTC Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) on a tablet computer.
quality of life (QoL) | Up to 5 years
  QoL measurement is additionally conducted in the hospital after treatment via digital questionnaire Functional Assessment of Cancer Therapy - Breast (FACT-B) on a tablet computer.

OTHER OUTCOMES:
Time from MRD turning positive until clinical relapse | Up to 5 years
  the mean time from MRD turning positive until clinical relapse
Coincidence rate between MRD continuing positive and clinical relapse | Up to 5 years
  the coincidence rate between MRD continuing positive and clinical relapse

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (3):
- China (3):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Huanxing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences, Hebei Center, Langfang, Hebei